CLINICAL TRIAL: NCT05644977
Title: A Phase 1, Randomized, Placebo-controlled Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Emraclidine Following Multiple Oral Doses in Healthy Elderly Participants (Part A) and to Evaluate the Safety and Tolerability of Emraclidine in Participants With Dementia Due to Alzheimer's Disease (Part B)
Brief Title: A Multiple Dose Trial of Emraclidine in Elderly Participants and in Participants With Dementia Due to Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CVL-231-1006
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants; Alzheimer's Disease Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Cohort 1: Emraclidine Dose 1 (Experimental): Participants will receive emraclidine dose 1 or emraclidine-matching placebo tablets, orally, once daily (QD) up to Day 14.
  Interventions: Drug: Emraclidine; Drug: Placebo
- Part A: Cohort 2: Emraclidine Dose 2 (Experimental): Participants will receive emraclidine dose 2 or emraclidine-matching placebo tablets, orally, QD up to Day 14.
  Interventions: Drug: Emraclidine; Drug: Placebo
- Part A: Cohort 3: Emraclidine Dose 3 (Experimental): Participants will receive emraclidine dose 3 or emraclidine-matching placebo tablets, orally, QD up to Day 14.
  Interventions: Drug: Emraclidine; Drug: Placebo
- Part A: Cohort 4: Emraclidine Dose 4 (Experimental): Participants will receive emraclidine dose 4 or emraclidine-matching placebo tablets, orally, QD up to Day 14.
  Interventions: Drug: Emraclidine; Drug: Placebo
- Part A: Cohort 5: Emraclidine Dose 5 (Experimental): Participants will receive emraclidine dose 5 or emraclidine-matching placebo tablets, orally, QD up to Day 14.
  Interventions: Drug: Emraclidine; Drug: Placebo
- Part B: Cohort 6: Emraclidine Dose 6 (Experimental): Participants with dementia due to AD will receive emraclidine dose 6 or emraclidine-matching placebo tablets, orally, QD up to Day 28.
  Interventions: Drug: Emraclidine; Drug: Placebo

INTERVENTIONS:
Drug: Emraclidine — Oral tablets
  Other Names: CVL-231; PF-06852231
Drug: Placebo — Oral tablets

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of emraclidine administered orally to healthy elderly participants in Part A (multiple ascending doses) and participants with dementia due to Alzheimer's disease (AD) in Part B.

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1 to 5 (Part A)

1. Male participants and female participants of nonchildbearing potential, ages 65 to 85 years, inclusive.
2. Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator.
3. Body mass index of 17.5 to 32.0 kilograms per square meter (kg/m^2), inclusive, and total body weight >45 kg (100 pounds [lb]) at Screening.
4. Female participants will be of nonchildbearing potential, defined as follows:

   • Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause, and confirmed with a serum follicle-stimulating hormone level >40 international units per milliliter (IU/mL).
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the full protocol.

Cohort 6 (Part B)

1. Male participants and female participants of nonchildbearing potential, ages 55 to 90 years, inclusive.
2. Have a clinical diagnosis of possible or probable Alzheimer's disease dementia according to the 2011 National Institute on Aging - Alzheimer's Association (NIA-AA) clinical criteria at the Screening Visit; diagnosis must be stable for at least 6 months prior to signing the ICF.
3. Have a Mini-Mental State Examination (MMSE) score of 8 through 26, inclusive, at the Screening Visit.
4. Have prior neuroimaging evidence (Computed Tomography [CT] or Magnetic resonance imaging [MRI] completed within the 3 years prior to signing the ICF) collected during or subsequent to the onset of dementia symptoms to rule out other central nervous system disorders that could account for the dementia syndrome.
5. Currently receiving oral symptomatic treatment for dementia (i.e., cholinesterase inhibitor and/or memantine), must have been on a stable regimen for at least 6 weeks prior to signing ICF and be willing to maintain a stable dose for the duration of the trial.
6. Body mass index of 17.5 to 40.0 kg/m2, inclusive, and total body weight >45 kg (100 lb) at Screening.

Exclusion Criteria:

All Cohorts

1. "Yes" responses for any of the following items on the C-SSRS (within the past 6 months):

   * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
   * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) "Yes" responses for any of the following items on the C-SSRS (within past 2 years):
   * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior). Serious risk of suicide in the opinion of the investigator is also exclusionary.
2. Diagnosis of moderate to severe substance or alcohol-use disorder (excluding nicotine or caffeine) as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria within 12 months prior to signing the ICF.
3. Positive drug screen or a positive test for alcohol at Screening or Baseline Visits.
4. Any of the following clinical laboratory test results at the Screening Visit (as assessed by the central laboratory) and at Check-in (Day -1; as assessed by the local laboratory), and confirmed by a single repeat measurement, if deemed necessary:

   * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.0 × upper limit normal (ULN)
   * Total bilirubin >1.5 × ULN. If Gilbert's syndrome is suspected, total bilirubin >1.5 × ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.

Cohorts 1 to 5 (Part A)

1. Current or past history of significant pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus), malignancy (except for basal cell carcinoma of the skin and cervical carcinoma in situ, at the discretion of the investigator), hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
2. Current or past history of significant cardiovascular disease.
3. Estimated glomerular filtration rate <60 milliliters per minute (mL/min)/1.73 m^2, as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI 2021) equation at the Screening Visit or Check-in (Day -1).

Cohort 6 (Part B)

1. Has either of the following:

   * History of major depressive episode with psychotic features during the 12 months prior to signing the ICF
   * History of a diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder
2. Has evidence of a clinically relevant neurological disorder other than possible or probable Alzheimer's disease such as, but not limited to, the following:

   * History of ischemic stroke within 12 months prior to signing the ICF or any evidence of hemorrhagic stroke
   * History of cerebral amyloid angiopathy, epilepsy, or central nervous system neoplasm
3. Estimated glomerular filtration rate <60 mL/min/1.73 m2, as calculated using the CKD-EPI 2021 equation the Screening Visit.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Day 28
Part A: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to Day 17
Part A: Number of Participants With Clinically Significant Changes in Laboratory Assessments | Up to Day 17
Part A: Number of Participants With Clinically Significant Changes in Vital Sign Measurements | Up to Day 17
Part A: Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 17
Part A: Changes in Suicidality Assessed Using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 17
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.
Part A: Number of Participants With Clinically Significant Findings in Extrapyramidal Symptoms Evaluated Using the Simpson Angus Scale (SAS) | Up to Day 14
  The SAS consists of a list of 10 symptoms of parkinsonism. Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms and a score of 4 representing a severe condition. The SAS total score is the sum of the scores for all 10 items.
Part A: Number of Participants With Clinically Significant Findings in Extrapyramidal Symptoms Evaluated Using the Abnormal Involuntary Movement Scale (AIMS) | Up to Day 14
  The AIMS assessment consists of 10 items describing symptoms of dyskinesia. Each item is rated on a 5-point scale, with a score of 0 representing absence of symptoms (for item 10, no awareness), and a score of 4 indicating a severe condition (for item 10, awareness, severe distress). In addition, the AIMS includes 2 yes/no questions that address the participant's dental status.
Part A: Number of Participants With Clinically Significant Findings in Extrapyramidal Symptoms Evaluated Using the Barnes Akathisia Rating Scale (BARS) | Up to Day 14
  The BARS consists of 4 items related to akathisia. The first 3 items are rated on a 4-point scale, with a score of 0 representing absence of symptoms and a score of 3 representing a severe condition. The global clinical evaluation is made on a 6-point scale, with a score of 0 representing absence of symptom and a score of 5 representing severe akathisia.
Part B: Number of Participants With TEAEs, Clinically Significant Changes in ECG Parameters, Laboratory Assessments, Vital Sign Measurements, and Physical and Neurological Examination Results | Up to Day 28
Part B: Changes in Suicidality Assessed Using the C-SSRS | Up to Day 28
Part B: Number of Participants With Clinically Significant Findings in Extrapyramidal Symptoms | Up to Day 28
  Extrapyramidal symptoms will be evaluated using SAS, AIMS, and BARS scales.

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of Emraclidine and its Metabolite CV-0000364 | Days 1 and 14
Part A: Time to Maximum Plasma Concentration (Tmax) of Emraclidine and its Metabolite CV-0000364 | Days 1 and 14
Part A: Area Under the Plasma Concentration-time Curve (AUC) of Emraclidine and its Metabolite CV-0000364 | Days 1 and 14
Part A: Trough Plasma Concentration (Ctrough) of Emraclidine and its Metabolite CV-0000364 | Days 1 and 14
Part A: Peak to Trough Ratio (PTR) of Emraclidine and its Metabolite CV-0000364 | Day 14
Part A: Apparent Clearance of Drug From Plasma (CL/F) of Emraclidine | Days 1 and 14
Part A: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Emraclidine | Days 1 and 14
Part A: Apparent Terminal Half-life (t1/2) of Emraclidine and its Metabolite CV-0000364 | Days 1 and 14
Part A: Accumulation Ratio (Rac) of Emraclidine and its Metabolite CV-0000364 | Day 14
  Rac would be calculated from AUC and Cmax of emraclidine and its metabolite.
Part A: Metabolite to Parent Ratio of Emraclidine and its Metabolite CV-0000364 | Days 1 and 14
Part B: Plasma Concentrations of Emraclidine and its Metabolite CV-0000364 | Days 1 to 28

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- United States (11):
  - Cypress, California, Cypress, California
  - San Diego, California, San Diego, California
  - Hialeah, Florida, Hialeah, Florida
  - Decatur, Georgia, Decatur, Georgia
  - Honolulu, Hawaii, Honolulu, Hawaii
  - Overland Park, Kansas, Overland Park, Kansas
  - Farmington Hills, Michigan, Farmington Hills, Michigan
  - Marlton, New Jersey, Marlton, New Jersey
  - Princeton, New Jersey, Princeton, New Jersey
  - Staten Island, New York, Staten Island, New York
  - North Canton, Ohio, North Canton, Ohio

IPD SHARING:
Plan to Share IPD: No